CLINICAL TRIAL: NCT03699254
Title: Efficacy and Safety of the Combination of Reduced Duration Prophylaxis Followed by Immuno-guided Prophylaxis to Prevent Cytomegalovirus Disease in Lung Transplant Recipients (CYTOCOR STUDY): An Open-label, Randomised, Non-inferiority Clinical Trial.
Brief Title: Clinical Trial of Efficacy and Safety of the Combination of Reduced Duration Prophylaxis Followed by Immuno-guided Prophylaxis in Lung Transplant Recipients.
Acronym: CYTOCOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYTOCOR; 2018-003300-39 (EudraCT Number)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Transplantation Infection; Cytomegalovirus Infections
Keywords: Lung transplantation; Cytomegalovirus infection; Specific immunity
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Control Group (universal prophylaxis + pre-emptive therapy; 6+6): The recommendation of the Spanish Consensus Document will be followed according to the strategy described below:
  * Universal prophylaxis with valganciclovir (900 mg/24h, corrected for renal function) up to month +6. The use of associated immunotherapy (e.g., anti-CMV hyperimmune immunoglobulin) will depend on each center's clinical practice. During this period, the treatment of blips of viral replication detected during the usual clinical follow-up of patients will depend oneach center's clinical practice.
  * Pre-emptive therapy guided by viral load from month +6 to month +12. For a viral load above> 38 copies/mL (> 35 IU/mL) and depending on each center's clinical practice, treatment with valganciclovir may be initiated (900 mg/12h, corrected for renal function).
  Interventions: Drug: Valganciclovir; Drug: Ganciclovir
- Experimental (Experimental): Experimental Group (reduced prophylaxis + immuno-guided prophylaxis; 3+9):
  * Universal prophylaxis with valganciclovir (900 mg/24h, corrected for renal function) up to month +3. The use of associated immunotherapy (e.g., anti-CMV hyperimmune immunoglobulin) will depend oneach center's clinical practice. During this period, the treatment of blips of viral replication detected during the usual clinical follow-up of the patients will depend on the each center's clinical practice.
  * Immuno-guided prophylaxis. This will consist of a monthly determination of cellular immunity by QF-CMV from month +3 to month +12.
  Interventions: Drug: Valganciclovir; Drug: Ganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir is a L-valyl ester of ganciclovir that exists as a mix of 2 diastereomers. After administration, both are converted to ganciclovir by esterases. Ganciclovir is a synthetic analogue of 2'-deoxyguanosine, it inhibits replication of cytomegalovirus.
  In CMV-infected cells it's phosphorylated (phosphorylation is dependent on the viral kinase and occurs preferentially in virus-infected cells). Ganciclovir activity is due to inhibition of viral DNA synthesis by ganciclovir triphosphate.
  Other Names: Valcyte
Drug: Ganciclovir — Ganciclovir is a synthetic analogue of 2'-deoxyguanosine, it inhibits replication of cytomegalovirus.
  In CMV-infected cells it's phosphorylated (phosphorylation is dependent on the viral kinase and occurs preferentially in virus-infected cells). Ganciclovir activity is due to inhibition of viral DNA synthesis by ganciclovir triphosphate.
  Other Names: Cymevene

SUMMARY:
To assess the efficacy of reduced duration prophylaxis followed by immuno-guided prophylaxis to prevent cytomegalovirus disease.

DETAILED DESCRIPTION:
Prolonged use of antivirals to prevent the development of cytomegalovirus (CMV) disease in lung transplant patients has been shown to have significant side effects, for which alternatives are being sought to reduce their use. The monitoring of cell immunity against CMV could be an alternative as it has shown to be useful in identifying transplant patients at low risk of infection, who could benefit from shorter prophylaxis. The aim of the CYTOCOR study is to demonstrate that the combination of a reduced prophylaxis strategy with subsequent CMV-specific immunological monitoring would allow CMV infection to be controlled in lung transplant patients as effectively as the usual strategy (prophylaxis followed by pre-emptive therapy), while reducing the side effects of antivirals due to the shorter duration of prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cytomegalovirus positive serology who underwent lung transplantation.
* Subjects of 18 years of age or older.
* Expected valgancilovir prophylactic treatment of 6 months after transplantation.
* Patients who have signed the informed consent form.

Exclusion Criteria:

* HIV infected subjects.
* Subjects unable to comply with the protocolo follow-up visits.
* Subjects who underwent multivisceral transplant.
* Pregnant and/or lactating women.
* Intolerance to Valganciclovir/Ganciclovir treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Cytomegalovirus disease incidence rate at 18 months after lung transplantation. | 18 months after subject's transplantation.
  Cytomegalovirus disease incidence rate at 18 months after lung transplantation.

SECONDARY OUTCOMES:
INFG cut-off point other than 0.2 IU/mL | 18 months after subject's transplantation.
  For patients of the experimental group (3+9) in which immuno-guided prophylaxis is used based on QF-CMV Reactive (cut-off 0.2 IU/mL of IFNG) and who develop CMV disease, a secondary objective will be to assess whether an INFG cut-off point other than 0.2 IU/mL could predict protection against the disease more reliably.

CONTACTS AND LOCATIONS:
Overall Officials: Julián de la Torre Cisneros, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (7):
- Spain (7):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Univesitario Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available.
  Individual parcicipant data that underlie the results reportes in this article, after deidenttification (text, tables, figures and appendices)
  The other documents that will be available: study protocol, Statistical Analysis Plan, Informed Consent Form.
  The data will be available beginning 9 months and ending 36 months following article publication.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Paez-Vega A, Vaquero-Barrios JM, Ruiz-Arabi E, Iturbe-Fernandez D, Alonso R, Ussetti-Gil P, Monforte V, Pastor A, Fernandez-Moreno R, Mora VM, Erro-Iribarren M, Quezada CA, Berastegui C, Cifrian-Martinez JM, Cano A, Caston JJ, Machuca I, Lobo-Acosta MA, Gutierrez-Gutierrez B, Cantisan S, Torre-Cisneros J; CYTOCOR study group. Safety and efficacy of immunoguided prophylaxis for cytomegalovirus disease in low-risk lung transplant recipients in Spain: a multicentre, open-label, randomised, phase 3, noninferiority trial. Lancet Reg Health Eur. 2025 Mar 26;52:101268. doi: 10.1016/j.lanepe.2025.101268. eCollection 2025 May. PMID 40224372
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Gibson L. An Interferon-gamma Release Assay for Evaluation of Cell-mediated Immunity in Infants With Congenital Cytomegalovirus Infection. Clin Infect Dis. 2021 Aug 2;73(3):374-375. doi: 10.1093/cid/ciaa700. No abstract available. PMID 32504089
- [Derived] Paez-Vega A, Cantisan S, Vaquero JM, Vidal E, Luque-Pineda A, Lobo-Acosta MA, Perez AB, Alonso-Moralejo R, Iturbe D, Monforte V, Otero-Gonzalez I, Pastor A, Ussetti P, Torre-Cisneros J. Efficacy and safety of the combination of reduced duration prophylaxis followed by immuno-guided prophylaxis to prevent cytomegalovirus disease in lung transplant recipients (CYTOCOR STUDY): an open-label, randomised, non-inferiority clinical trial. BMJ Open. 2019 Aug 15;9(8):e030648. doi: 10.1136/bmjopen-2019-030648. PMID 31420397